CLINICAL TRIAL: NCT00912704
Title: Prevention and Treatment of Chronic Kidney Disease in Taiwan - Development of Early Diagnostic Techniques and Setup of Local Therapeutic Guidelines and Standards
Brief Title: Development of Early Diagnostic Techniques and Setup of Local Therapeutic Guidelines and Standards
Acronym: Hmodialysis
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Collaborators: Wake Forest University Health Sciences (Other)
Responsible Party: Far Eastern Memorial Hospital, Hospital
Other Study IDs: 098001-3
Record Dates: First submitted 2009-06-02; First posted 2009-06-03 (Estimated); Last update posted 2009-06-03 (Estimated); Status verified 1998-04

CONDITIONS: Healthy
Keywords: Hemodialysis patients; Kidney; Physician attitudes; Family wishes; 30 numbers require maximum

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
End-stage renal disease (ESRD) is a healthy, social and economic threat worldwide. In the past ten years, the incidence and prevalence of ESRD patients have tremendously increased, ranking at the top in the world. The reasons for such high incidence and prevalence are multifactor. Early diagnosis and closed monitor of the patients with chronic kidney disease (CKD) may be beneficial, but not confirmed yet.The advising mechanisms for non-doing or withdraw long-term dialysis. All these studies will be performed in a multicentered project. Three medical centers in which CKD researches have been conducted for many years will provide a large cohort and share the data collected from their own hospitals. We expect that the results will provide an excellent guideline for CKD care, achieve cost-effectiveness of dialysis therapy and better life quality of ESRD patients.

DETAILED DESCRIPTION:
Purpose: Development of early diagnostic techniques and setup of local therapeutic guidelines and standards.

Design: The group plans to host the co-operation of hospitals, based on the geographical distribution of co-operation of several hospitals to choose the renal physician interviews the doctor and patient received a total of 30 objects was conducted qualitative in-depth interviews.

Time:2008/9/1~2011/8/31

Inclusion criteria): To withdraw from dialysis treatment of chronic kidney disease, qualitative research, to-depth interviews, field observation, video recording, and public hospitals at the same time the collection of literature.

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease patients with the end of dialysis to withdrawal.

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Not limited to the patient himself, as soon as the patient or family members decide to enter or removed after dialysis can be done by patients themselves or family members as well as the main decision-depth interviews with relevant medical and nursing staff.
  Recently, a relative of reference are as follows:
  1. Spouse.
  2. Adult direct blood relatives of British Columbia.
  3. Parents.
  4. Brothers and sisters.
  5. Grandparents.
  6. Three pro-grandparents or extended family, such as blood.
  7. Pro-marriage and so immediate.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 1998-03; Primary Completion 1998-03 (Actual); Study Completion 1998-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chang Duan-Rong, doctor, Principal Investigator — the Institute of Health Care Organization Administration (IHCOA)